CLINICAL TRIAL: NCT00842491
Title: A Phase II Study of Endostar (Recombinant Human Endostatin ®) With Cisplatin and Capecitabine (Xeloda) as 1st Line Treatment in the Advanced Gastric Cancer
Brief Title: Study of Endostar With Cisplatin and Capecitabine as 1st Line Treatment in the Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Xiansheng Pharmaceutical Company (Unknown)
Responsible Party: Principal Investigator, Shen Lin, pro., Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDOCX
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — endostar protein; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- endostar+chemotherapy (Experimental)
  Interventions: Drug: endostar, cisplatin, capecitabine; Drug: capecitabine; Drug: cisplatin

INTERVENTIONS:
Drug: endostar, cisplatin, capecitabine — Product 1: endostar
  Dosing schedule: 15mg daily dose, d1-14
  Mode of administration: intravenously
Drug: capecitabine — Product 2: capecitabine
  Dosing schedule: 1000mg/m2 bid, days 1-14, every 3 weeks
  Mode of administration: orally
Drug: cisplatin — Product 3: cisplatin
  Dosing schedule: 80mg/m2, day 1 of every 3 weeks
  Mode of administration: intravenously

SUMMARY:
The purpose of this study is to investigate whether endostar (recombinant human endostatin)with cisplatin and capecitabine (Xeloda) as 1st line treatment in the advanced gastric cancer is effective and safe.

DETAILED DESCRIPTION:
Endostar, a recombinant human endostatin, has shown its antitumor ability in combination in NSCLC and breast cancer. But to gastric cancer, few clinical data has been reported. However, bevacizumab, an angiogenesis inhibitor was shown effective in combination with chemotherapy in advanced gastric cancer in some phase II study. So in this study, we want to explore whether endostar is also effective and safe in advanced gastric cancer. Response predictive factor is expected to be identified.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age 18 to 70 years old
* Histologically confirmed gastric adenocarcinoma
* Unresectable recurrent or metastatic disease
* Previous neo-adjuvant or adjuvant treatment for gastric cancer, if applicable, more than 6 months
* Previous chemotherapy with capecitabine or cisplatin, if applicable, more than 12 months.
* Measurable disease according to the RECIST criteria
* Karnofsky performance status ≥60
* Life expectancy of ≥2 month
* No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)
* Serum albumin level ≥3.0g/dL
* Serum AKP < 2.5 times ULN
* Serum creatinine <ULN, and CCr < 60ml/min
* Bilirubin level < 1.5 ULN
* WBC>3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Brain metastasis (known or suspected)
* Previous systemic therapy for metastatic gastric cancer
* Inability to take oral medication
* Previous therapy targeting at angiogenesis or vasculogenesis pathway or other targeted therapy
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry
* Contraindications of nuclear magnetic resonance image such as fitment of cardiac pacemaker , nerve stimulator, or aneurysm clip, and metallic foreign body in eye ball and so on.
* Allergic constitution or allergic history to protium biologic product or any investigating agents.
* Severe heart disease or such history as recorded congestive heart failure, uncontrolled cardiac arrhythmia, angina pectoris needing medication, cardiac valve disease, severe abnormal ECG findings, cardiac infarction , or retractable hypertension.
* Pregnancy or lactation period
* Any investigational agent within the past 28 days
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Previous adjuvant therapy with capecitabine+platinum,
* Pre-existing neuropathy>grade 1
* Legal incapacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 year

SECONDARY OUTCOMES:
Tumor response rate | 1 year
Disease control rate | 1 year
Overall survival | 5 year
adverse evens | 5 year
The alteration of relative regional blood volume of the tumor | 3weeks

CONTACTS AND LOCATIONS:
Overall Officials: lin shen, MD, Principal Investigator — Peking University, School of oncology, Department of GI oncology
Locations (1):
- Department of GI Oncology, Peking University, School of Oncology, Beijing, Beijing Municipality, China